#### University of Minnesota Bone Marrow Transplantation Program

# MT2005-21 AUTOLOGOUS PERIPHERAL BLOOD STEM CELL TRANSPLANT FOR GERM CELL TUMORS VERSION 4

Principal Investigator: Najla El Jurdi, MD

Co-Investigators: Claudio Brunstein, MD, PhD Daniel Weisdorf, MD Jeffrey S. Miller, MD Todd Defor, MS (Statistician)

July 12, 2019

#### TABLE OF CONTENTS

| SCHEMA | Р4 |
|---|---|
| 1.0 BACKGROUND AND RATIONALE | P6 |
| 2.0 Objectives | |
| 3.0 ELIGIBILITY AND EXCLUSION CRITERIA | |
| 4.0 Subject Registration. | р11 |
| 5.0 Treatment Plan | Р12 |
| 6.0 Required Observations. | Р16 |
| 7.0 Transplant related Toxicities and Complications | Р17 |
| 8.0 Adverse Event Reporting | Р20 |
| 9.0 Data and Safety Monitoring | Р21 |
| 10.0 Experimental Design and Statistical Considerations | Р22 |
| 10.0 RETENTION OF RECORDS. | Р23 |
| 11.0 References. | P23 |
| APPENDICIES APPENDIX I: INTERNATIONAL GERM CELL CANCER CONSENSUS CLASSIFICATION APPENDIX II: KARNOFSKY AND LANSKY PERFORMANCE SCALE APPENDIX III: REQUIRED OBSERVATIONS APPENDIX IV: RECIST CRITERIA FOR MEASUREMENT OF DISEASE RESPONSE | |
| APPENDIA IV. RECISI CRITERIA FOR MIEASUREMENT OF DISEASE RESPONSE | |

#### **PI Contact Information:**

Najla El Jurdi, MD Division of Hematology/Oncology/Transplantation MMC 480 420 Delaware Street SE Minneapolis, MN 55455 612 625-8942 (phone) neljurdi@umn.edu (email)

## **Revision History**

| Date | Revision details | Consent change/<br>version date |
|---|---|---|
| 1-29-07 | The goal collection is 10 X 10 <sup>6</sup> CD34 <sup>+</sup> cells/kg instead of 6 X 10 <sup>6</sup> CD34 <sup>+</sup> cells/kg to reflect a goal of 5 x10 <sup>6</sup> CD34 <sup>+</sup> cells/kg for infusion for each transplant. | |
| 3-13-2008 | Clarified exclusion criteria to state that patients with progressive disease will not be eligible for a second transplant, added RECIST criteria (as appendix IV), fixed typo in section 5.5 | |
| | Removed Dr. Nasfat Shehadeh from protocol team | |
| 6-15-09 | Dr. Brian McClune takes over as PI; Dr Tomblyn removed from study | |
| 9/9/2009 | Typo correction in schema | |
| 9/27/2010 | Typo correction in schema | |
| 1/10/11 | Error correction in peds fluid hydration rate | |
| 09/12/2018 | Dr Brunstein is PI | |
| 07/12/2019 | Dr. El Jurdi takes over as Principal Investigator | Y |

#### **SCHEMA**

#### MOBILIZATION AND STEM CELL COLLECTION



#### **TRANSPLANT**

#### Admit within 2 weeks of completing Cell Collection



Standard transplant follow-up (see appendix IIIB)

#### 1.0 Background And Rationale

#### 1.1 BACKGROUND

Germ cell tumors (GCT) are highly sensitive to chemotherapy such that even with metastatic disease at diagnosis, many patients can be cured—greater than 90% 5-year overall survival—at the time of diagnosis<sup>1</sup>. The International Germ Cell Consensus Classification divides patients based on risk factors into good, intermediate and poor prognostic categories to better estimate outcomes [Appendix I]<sup>2</sup>. Many patients who fall into the poor risk category or other patients who relapse are successfully salvaged with high dose chemotherapy and autologous stem cell transplant (AuSCT)<sup>3-6</sup>.

Beyer and colleagues analyzed 310 patients at four institutions to determine prognostic factors in patients with relapsed GCT treated with AuSCT<sup>7</sup>. Four factors were found to be important in multivariate analysis (Beyer Index):

- progressive disease after salvage therapy immediately prior to transplant
- absolute cisplatin refractory disease (defined as progressive increase in serum markers despite on-going cisplatin chemotherapy) or cisplatin refractory disease (defined as disease progression within 4 weeks of a the last cycle of chemotherapy)
- an hCG level of > 1000 IU/L
- primary mediastinal non-seminomatous GCT

Patients with more than 2 of these factors were considered poor risk with a 2 year relapse free survival of only 5% versus 51% for patients with no risk factors and 27% in patients with 1 or 2 risk factors.

There are other diseases, such as myeloma, in which sequential high dose chemotherapy and AuSCT have demonstrated improved overall and disease free survival<sup>8</sup>. Prior investigations in GCT suggest that a subset of high risk or relapsed patients may be cured with sequential cycles of high dose chemotherapy and AuSCT<sup>4,9</sup>. Interestingly, in the initial prognostic study by Beyer, only 20% of patients were treated with two transplants. An initial pilot study from Margolin et al, demonstrated feasibility of tandem high-dose chemotherapy with AuSCT in a cohort of patients with either high-risk primary disease in partial response or platinum-sensitive relapse<sup>9</sup>. Both conditioning cycles consisted of ifosfamide, carboplatin, and etoposide (ICE). Treatment related mortality was zero and at almost 4 years, 9 of 20 patients enrolled were alive and disease-free. Other studies have looked at sequential therapy with regimens including paclitaxel, a drug found effective in cisplatin-refractory patients<sup>10</sup>. A recent study utilized paclitaxel in both conditioning regimens in 33 patients<sup>11</sup>. At a median follow-up of 5 years, 36% of patients were

alive without disease although only 2 (18%) patients with a Beyer index of  $\geq$  2 remained progression-free after therapy. Table 1 gives a summary of several studies investigating AuSCT for GCT.

#### 1.2 RATIONALE

The use of either non-cross resistant therapy or more than two high dose therapy cycles are areas of interest<sup>4,10</sup>. In this study, we propose to use tandem transplant with non-cross resistant conditioning regimens to further study these issues. Pre clinical and clinical studies have found that taxanes can salvage patients with cisplatin-refractory GCT<sup>10-14</sup>. As documented in Table 1, most prior studies have not used non-cross resistant conditioning regimens for AuSCT but rather identical conditioning for both transplants. We propose that patients with high-risk or relapsed disease may benefit from using chemotherapeutic agents that have differing mechanisms of action and differing resistance patterns as high dose therapy. This would permit tumor kill prior to development of further resistance.

Mobilization of sufficient numbers of peripheral blood stem cells may not occur in all patients. For those patients collecting  $\geq 2 \times 10^6$  CD34<sup>+</sup> cells/kg but  $< 4 \times 10^6$  CD34<sup>+</sup> cells/kg, only a single transplant can safely be performed. However, it would be inappropriate to deny them AuSCT which is a demonstrated salvage regimen with potential for cure. This protocol accounts for this possibility by providing a treatment option for patients with insufficient PBSC collection for tandem transplantation. The conditioning regimen for the single transplant is identical to the conditioning regimen of Transplant 1 for planned tandem patients.

Table 1

| Author | Study Type | Treatment | Patients | N | Response | EFS | OS |
|---|---|---|---|---|---|---|---|
| Vaena <sup>15</sup> | Retrospective | Carbo + VP16 conditioning;<br>tandem AuSCT if possible | Relapsed, cisplatinum refractory | 80 (56 received x2 AuSCT) | 45% | 32% (2y) | 40% (2y) |
| Rick <sup>16</sup> | Phase II | TIP x3 then Carbo+VP16+TT conditioning | Relapsed disease | 80 (62 SCT) | 78% (of patients transplanted) | 25% (3y) | 30% (3y) |
| Motzer <sup>10</sup> | Phase I/II | Paclitaxel + Ifos x 2 then<br>Carbo + VP16 conditioning | Relapsed cisplatinum<br>refractory and poor<br>prognostic features | 37 | 62% | 49% (31 months) | 54% (31<br>months) |
| Motzer <sup>17</sup> | Phase II | Carbo + VP16 + Cy; tandem<br>AuSCT if possible | Relapsed/refractory disease | 58 (27 received x2 AuSCT) | 40% CR | 21% (2y) | 31% (2y) |
| Bhatia <sup>3</sup> | Retrospective | Carbo + VP16 x2 | Relapsed/refractory disease | 65 (58 received x2 AuSCT) | 63% CR | 57% (3y) | 68% (3y) |
| Nichols <sup>6</sup> | Phase II (multicenter) | Carbo + VP16; x2 if possible | Relapsed or refractory disease | 38 (22 received x2 AuSCT) | 45%<br>(24% CR) | 13% (1y) | 35% (1y) |
| Mandanas <sup>5</sup> | Retrospective | Cy + Carbo + VP16 (68% of patients) | Relapsed or refractory | 21 (1 received x2 AuSCT) | 79% | 52% (3y) | 52% (3y) |
| Lotz <sup>4</sup> | Phase II<br>(multicenter) | Epi + Paclitaxel x2 then TT<br>+CY conditiong for SCT1<br>then ICE conditioning for<br>SCT 2 and 3 | Relapsed, poor prognosis disease | 45 (7 received x2 SCT, 22 x3 SCT) | 38% | 24% (3y) | 24% (3y) |
| Rosti <sup>18</sup> | Retrospective | Carbo + VP16 (19); ICE<br>(30); Carbo + VP16 + CY<br>(35) | Relapsed disease | 84 (19 received x2 SCT, 1 x 3 SCT) | 45% CR | 30% (5y) | 33% (5y) |
| Margolin <sup>9</sup> | Phase I/II | ICE conditioning; tandem<br>AuSCT | Poor prognosis,<br>chemotherapy<br>sensitive disease | 20 (18 received x2 AuSCT) | 60% | 45% (3y) | 45% (3y) |
| Margolin <sup>11</sup> | Phase I/II | Paclitaxel + Carbo + VP16<br>(SCT1); Paclitaxel + Carbo +<br>Ifosfamide (SCT2) | Relapsed or refractory GCT | 33 (2 received no SCT; 19 received x2 AuSCT) | Not reported | 36% (5y) | 42% (5y) |

Carbo = carboplatinum, VP16 = etoposide, TT = thiotepa, Cy = cyclophosphamide, Epi = epirubicin, ICE = Ifosfamide + Carboplatinum + Etoposide EFS = Event-free survival, OS = overall survival, Response = CR + PR unless otherwise stated

7/12/2019 

#### 2.0 Objectives

End organ toxicities such as myelosuppression often dictate the maximal doses of chemotherapy that can be administered safely. Autologous peripheral blood stem cell transplant (AuSCT) after high-dose chemotherapy circumvents this marrow toxicity allowing for dose intensification. This has been demonstrated to be useful in the salvage setting for patients with relapsed germ cell tumor (GCT)<sup>3-6</sup> The use of non-cross resistant chemotherapy regimens should increase the overall and disease-free survival in patients with high risk or relapsed GCT.

#### 2.1 Primary Objective

To determine overall survival for patients with GCT treated with tandem AuSCT with non-cross-resistant conditioning regimens.

#### 2.2 Secondary Objectives

- 2.2.1 To determine disease-free survival for patients with GCT treated with tandem AuSCT with non-cross-resistant conditioning regimens
- 2.2.2 Evaluate toxicity of tandem AuSCT
- 2.2.3 Evaluate time to engraftment of neutrophils and platelets for each transplant
- 2.2.4 Determine numbers of patients unable to adequately mobilize sufficient peripheral blood stem cells (PBSC) for tandem transplant
- 2.2.5 Identify prognostic factors of those patients unlikely to mobilize sufficient PBSC for tandem transplant
- 2.2.6 Compare outcomes of overall and disease free survival for patients undergoing single versus tandem transplant due to biologic randomization

#### 3 Eligibility Criteria

- 3.1 Diagnosis: Poor Prognosis Non-Seminomas Germ Cell Tumor in ≥ PR1/CR1 or Good or Intermediate Prognosis Seminomas and Non-Seminomas Germ Cell Tumor in ≥ PR1 or ≥ CR2 as defined by the International Germ Cell Cancer Consensus Classification (appendix I) Patients with increasing tumor markers only (i.e. no imaging evidence of progressive disease) are eligible for transplant.
- 3.2 Age:  $\geq 10$  years and  $\leq 70$  years of age.
- 3.2 Performance status: Karnofsky  $\geq 80\%$  (subjects  $\geq 16$  years of age) Lansky  $\geq 80\%$  for subject 10 - 15 years of age [Appendix II]
- **3.3 Life expectancy:** Greater than 8 weeks.

- **3.4** Patients must have normal organ function as defined below:
  - 3.4.1 Hematologic:

Hemoglobin > 8 gm/dL without transfusion and off erythropoietin for 14 days or Aranesp for 21 days

WBC > 2.5 x  $10^9$ /L with an ANC > 1.5 x  $10^9$ /L and off G-CSF or GM-CSF for 10 days or Neulasta for 21 days

Platelets  $> 100 \times 10^9$ /L without transfusion and/or a bone marrow cellularity of  $\ge 20\%$ 

- 3.4.2 Renal: Creatinine  $\leq 2.0$  mg/dl or creatinine clearance  $\geq 50$  ml/min.
- 3.4.3 <u>Hepatic:</u> Total bilirubin ≤ 2.0 mg/dl, AST and alkaline phosphatase < 5 x upper limit of normal. No history of severe prior or ongoing chronic liver disease.
- 3.4.4 <u>Cardiac</u>: Patients must be free of symptoms of uncontrolled cardiac disease including unstable angina, decompensated congestive heart failure, or arrhythmia. LVEF ≥45% by MUGA/ECHO
- 3.4.5 <u>Pulmonary:</u> Patients must have no significant obstructive airways disease (FEV<sub>1</sub> must be  $\geq$  50% of predicted) and must have acceptable diffusion capacity (corrected DLCO > 50% of predicted).
- 3.5 Patients with a history of CNS tumor involvement are eligible if they have completed treatment for CNS disease (radiotherapy or surgery or chemotherapy), have recovered from or stabilization of the side effects associated with the therapy and have no evidence of progressive CNS disease at the time of enrollment
- **3.6** Patients with serious uncontrolled infections will not be eligible.
- 3.7 Male and female patients of reproductive potential must use an approved contraceptive method if appropriate (for example, intrauterine device [IUD], birth control pills, or barrier device) during and for the duration of study participation. The drugs used in this study are pregnancy category D clear evidence of risk in pregnancy. Pregnant and breast feeding women will not be eligible.
- 3.8 Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

- **3.9** Additional Eligibility prior to Transplant Two
  - 3.9.1 Total Collection of  $\geq$  4 x 10<sup>6</sup> CD34 cells/kg prior to transplant one
  - 3.9.2 Transplant able to occur between day +30 and day +90 from transplant one
  - 3.9.3 Recovery of blood counts as demonstrated by: WBC >  $2.5 \times 10^9$ /L with an ANC >  $1.5 \times 10^9$ /L and off G-CSF for 3 days
    Platelets >  $50 \times 10^9$ /L without transfusion in the prior 7 days
  - 3.9.4 Renal: Creatinine  $\leq 2.0 \text{ mg/dl}$  or creatinine clearance  $\geq 50 \text{ ml/min}$
  - 3.9.5 <u>Hepatic</u>: Total bilirubin  $\leq$  2.0 mg/dl, AST and alkaline phosphatase  $\leq$  5 x upper limit of normal
  - 3.9.6 <u>Infection:</u> Patients with serious uncontrolled infections at the time of planned transplant will be excluded
  - 3.9.7 Patients with progressive disease by RECIST criteria (Appendix IV) by imaging techniques are not eligible to proceed to the second transplant. Tumor marker increase alone is not sufficient to diagnose disease progression.

#### 4 Subject Registration

Informed consent must be signed prior to the performance of any study related procedures or assessments.

To be eligible for registration to this study, the patient must meet each criteria listed on the eligibility checklist based on the eligibility assessment documented in the patient's medical record. No exemptions or waivers will be granted for patients who do not meet the eligibility criteria.

#### 4.1 Registration with the University of Minnesota Clinical Trials Office (CTO)

To register a patient to this study, complete the Subject Registration Form and study specific eligibility checklist and fax it to the Clinical Trials Office Registrar at (612) 625-3624. Confirmation of registration with the study assigned patient ID number will be returned by email and/or fax within 1 working day.

#### 4.2 Patients who are registered and do not begin study treatment

If a patient is registered to the study, and is later found not able to begin the planned study treatment, for whatever reason, the patient will be removed from study and treated at the physician's discretion. The CTO Registrar will be notified of the patient's non-treatment status. Study data will be collected until the time the patient is off study. The reason for removal from study will be clearly indicated on the case report forms. The registration number cannot be reassigned.

#### 5 TREATMENT PLAN

#### 5.1 G-CSF Mobilization of Peripheral Blood Hematopoietic Stem Cells

Patients will be treated with Granulocyte colony stimulating factor (G-CSF)  $10\mu g/kg/day$  (rounded to the nearest vial size) beginning 5 days before the first planned apheresis and continuing until the last aphereresis.

Begin peripheral blood stem cell collection per section 5.2 on day 5 of G-CSF mobilization.

#### 5.2 Peripheral blood stem cell collection

Daily peripheral blood stem cell collection will continue for a minimum of 3 days unless the goal of  $10 \times 10^6$  CD34<sup>+</sup>/kg is reached earlier.

#### Minimum collection criteria for continuing collection:

The first collection must yield  $\geq 0.1 \times 10^6$  CD34 cells/kg After the second collection a total of  $\geq 0.3 \times 10^6$  CD34 cells/kg must have been collected. If either of these conditions is not met, apheresis is discontinued and the subject will begin Chemotherapy Mobilization per section 5.3.

#### Total cell collection of $\geq 4 \times 10^6 \text{ CD34}^+ \text{ cells/kg}$

A total cell collection of  $\geq 4 \times 10^6$  CD34<sup>+</sup> cells/kg is considered sufficient for the tandem transplant (Transplant 1 plus Transplant 2). The collected PBSC will be cryopreserved such that approximately 50% of the leukapheresed product can be thawed and infused for each transplant. Patient will proceed to transplant 1 per section 5.4.

# Total cell collection of $\geq 2 \times 10^6 \text{ CD34}^+$ cells/kg but $\leq 4 \times 10^6 \text{ CD34}^+$ cells/kg

If patients cannot be adequately collected with GCSF mobilization ( $< 4 \times 10^6$  CD34<sup>+</sup> cells/kg) Chemotherapy Mobilization will be done per section 5.3.

**5.3 Chemotherapy Mobilization and cell collection** (for patients with a total cell collection of  $< 4 \times 10^6 \text{ CD34}^+ \text{ cells/kg}$ )

#### **Chemotherapy mobilization:**

Mesna 800mg/m<sup>2</sup> IV

Cyclophosphamide 4gm/m<sup>2</sup> intravenously (IV) over 2 hours

**Mesna** 800mg/m<sup>2</sup> IV 3 hours, 6 hours, 9 hours, and 12 hours following the cyclophosphamide

G-CSF 10µg/kg/day (rounded to nearest vial size) beginning 72 hours after completion of cyclophosphamide (day 4) and continuing until leukapheresis is completed

The dose of cyclophosphamide will be calculated using actual body weight unless the patient is ≥120% of Ideal Body Weight (IBW) in which case, the Cyclophosphamide dose will be based on Adjusted Ideal Body Weight (AIBW).

 $IBW_{men} = 50kg + 2.3kg$  (inches of height over 60in)  $IBW_{women} = 45kg + 2.3kg$  (inches of height over 60in)

AIBW = IBW + 1/3(ABW - IBW)

Standard Cyclophosphamide hydration orders will be used.

Monitor CBC daily starting on day 4. Leukapheresis will start on the first day following an absolute neutrophils count (ANC)  $\geq 700/\mu L$ .

#### Minimum collection criteria for continuing collection:

The first collection must yield  $\geq 0.1 \times 10^6$  CD34 cells/kg After the second collection a total of  $\geq 0.3 \times 10^6$  CD34 cells/kg must have been collected.

If patient has received chemotherapy mobilization and the minimum criteria cannot be met, the cell collection should be stopped. If the patient has collected  $> 2 \times 10^6$  CD34 cells/kg with the combined aphereses, the patient is eligible for a single transplant. If the total collections are  $< 2 \times 10^6$  CD34 cells/kg, the patient is removed from study, and other treatment options discussed.

#### 5.4 Transplant One

Admit for transplant within two weeks of completing cell collection.

| Day | Drug | Administration |
|---|---|---|
| -8 (Admit) | | Admit to start premedications per section 5.4.1 and |
| | | hydration per section 5.4.2 |
| - 7 | Paclitaxel | 225 mg/m <sup>2</sup> IV over 3 hours starting at 0900 |
| | | • Dilute in 5% dextrose or 0.9% saline to a |
| | | concentration of 0.3 – 1.2 mg/mL |
| | | • Administer using a 0.22μM filter and polyethylene- |
| | | lined administration set |
| -6, -5, -4 | Ifosfamide | 2500mg/m²/day continuous infusion IV starting at 0900 |
| | Mesna | 2500mg/m <sup>2</sup> /day continuous infusion IV starting at 0900 |
| | | • See section 5.4.3 for ifosfamide dose calculation |
| | | • Combine mesna and ifosfamide in 1L D <sub>5</sub> W |
| 0 | | PBSC infusion |
| +5 until ANC ≥ | G-CSF | 5μg/kg/day (round to nearest vial size) SC or IV. May |
| 1500/μL for 3 | | be restarted if ANC falls below 1000/μL |
| consecutive days | | · |

#### 5.4.1 Premedication for Paclitaxel administration

- <u>Dexamethasone</u> 20 mg PO at 12 hours and 6 hours before administration. For pediatric patients, 5 mg/m<sup>2</sup> q 12 hrs
- <u>Diphenhydramine</u> 50mg IV 30 minutes before administration. For pediatric patients, 1 mg/kg q 6 hrs
- Ranitidine 50mg IV 30 minutes before administration. For pediatric patients, 1-2 mg/kg/day divided q 8 hrs

#### 5.4.2 Hydration

Normal Saline at 100mL/hour starting 10 hours before paclitaxel administration. For pediatric patients, slower infusion rates may be used with a goal infusion of 1500 ml/m<sup>2</sup> over 24 hours

At the completion of paclitaxel infusion, hydration should be increased to  $2000 - 3000 \text{ mL/m}^2/\text{day}$  until 24 hours after completion of ifosfamide.

Adequate diuretics should be given and patients urged to urinate every 1 - 2 hours to ensure urinary output of at least 200 mL every 2 hours and to maintain appropriate fluid balance. Patients should

be weighed BID during ifosfamide administrations to aid in managing fluid balance.

#### **5.4.3** Dosing of Ifosfamide

Dosing of ifosfamide will be per actual body weight unless the patient is ≥120% of Ideal Body Weight (IBW) in which case, the Ifosfamide dose will be based on Adjusted Ideal Body Weight (AIBW)

$$IBW_{men} = 50 \text{ kg} + 2.3 \text{kg}$$
 (inches of height over 60in)  
 $IBW_{women} = 45 \text{ kg} + 2.3 \text{kg}$  (inches of height over 60in)

$$AIBW = IBW + 1/3(ABW - IBW)$$

For patients qualifying to have only a single transplant (due to a collection of  $< 4 \times 10^6 \text{ CD34}^+ \text{ cells/kg}$ ) follow-up will be per appendix IIIA.

For patients qualifying to have a tandem transplant (transplant one and transplant two), study participation will continue per section 5.5.

#### 5.5 Transplant Two

Admission for transplant two will be no earlier than day 30 from first transplant and no later than day 90. Goal for admission is day 40-60. See section 3.9 for additional eligibility criteria for continuing with transplant 2.

| Day | Drug | Administration |
|---|---|---|
| -7 (Admit) | | Admit to start hydration per section 5.5.1 |
| -6, -5, -4 | Carboplatin | 500mg/m <sup>2</sup> /day IV over 60 minutes |
| -6, -5, -4 | Thiotepa | 150mg/m <sup>2</sup> /day IV over 30 minutes; see section 5.5.2 |
| | | for skin care |
| -6, -5, -4, -3 | Etoposide | 600mg/m <sup>2</sup> /day IV over 60 minutes |
| 0 | | PBSC infusion |
| +5 until ANC | G-CSF | 5μg/kg/day (round to nearest vial size) SC or IV. May |
| $\geq 1500/\mu L$ for | | be restarted if ANC falls below 1000/μL |
| 3 consecutive | | |
| days | | |

#### 5.5.1 Hydration

0.45% saline at 100mL/hour starting 10 hours before chemotherapy administration.

<u>For pediatric patients</u>, slower infusion rates may be used with a goal infusion of 1500ml/m<sup>2</sup> over 24 hours

#### 5.5.2 Thiotepa

Because Thiotepa can be excreted through the skin, the following precautions should be followed until 24 hours after the last dose is given:

- Beginning 3 4 hours after the first dose, bathing with soap and water should be done 3 – 5 times per day and pat dry to avoid skin irritation.
- Change lines, clothes, and central line dressing after each bath
- Avoid moisturizer, barrier creams, antiperspirants, and deodorants during treatment

#### 6 Required Observations (Appendix III A and III B)

- **6.1** Required observations are listed in Appendix III. The required observations for Transplant 1 (Appendix IIIA) will continue until 2 weeks before admission for Transplant 2 (Appendix IIIB).
  - 6.1.1 If the patient is not eligible to move forward to Transplant 2 (see section 3.11) then all required observations for Transplant 1 will continue.
  - 6.1.2 If the patient is eligible for Transplant 2 between day +30 and day +90, then the required observations for Transplant 2 will become effective at the time eligibility is determined. If the patient has had investigations performed (i.e. serum tumor markers on day +42) within the 2 weeks prior to admission for Transplant 2 (day +50 scheduled admission), these will not need repeated and the values obtained from the Transplant 1 observations will be used.
- **6.2** Staging studies prior to enrollment to define the extent of disease will include unilateral bone marrow aspiration and bilateral bone marrow biopsy, PET/CT scans of chest, abdomen, pelvis and brain, serum tumor markers including AFP, β-hCG, and LDH
  - If patient has had <u>no prior bone marrow involvement</u>, then bone marrow biopsies will be performed to determine eligibility and then at yearly intervals unless otherwise clinically indicated.
- **6.3** Imaging will be performed prior to enrollment in study; at Day +28, at Day +100, at Day +180, at 1 year and then at 6 month intervals in the second post-transplant year. Day +28 staging will be with a CT scan only. All other imaging will be with a PET/CT.
- **6.4** Serum tumor markers including AFP, β-hCG, and LDH will be checked every 2 weeks from transplant until day+100 and then at 6, 9, and 12 months post

transplant. After 1 year, tumor markers will be checked every 6 months until 2 years post-transplant.

### 7 Transplant Related Toxicities and Complications

#### 7.1 G-CSF mobilization:

| Frequency | Toxicity |
|-----------|------------------------------------|
| Common | Bone or muscle aches |
| | • Fever or chills |
| | • Discomfort at the injection site |
| | Malaise |
| Uncommon | • Skin rash |
| | Headache |
| Rare | Polyserositis |

#### 7.2 Peripheral blood stem cell collections

| Frequency | Toxicity |
|-----------|-------------------------------------------------------|
| Common | Mild discomfort at the site of catheter placement |
| Uncommon | Hypotension |
| | Thrombocytopenia might develop transiently following |
| | the leukopheresis and, if necessary, irradiated Blood |
| | Bank platelet concentrates will be transfused. |

#### 7.3 Chemotherapy Mobilization:

| | Cyclophosphamide (Cytoxan) |
|---|---|
| Frequency | Toxicity |
| Common | <ul> <li>Nausea and vomiting (aggressive anti-emetic therapy may minimize)</li> <li>Diarrhea</li> </ul> |
| | <ul> <li>Alopecia usually reversible, but changes in hair color or<br/>texture after regrowth may occur</li> </ul> |
| | <ul> <li>Permanent sterility is likely at this dose of<br/>cyclophosphamide, particularly when given with other<br/>drugs</li> </ul> |
| Uncommon | • Skin rash |
| | • Hemorrhagic cystitis may occur following the use of cyclophosphamide despite aggressive fluid replacement, frequent voiding and Mesna |

| Rare | • Pericarditis |
|------|------------------------------------------------------------|
| | • Cardiomyopathy: cyclophosphamide can cause fatal |
| | cardiac necrosis with clinical irreversible heart failure. |
| | • EKG changes are not infrequent and reduction in EKG |
| | voltage may be observed. Patients with compromised |
| | ejection fraction, previously treated with anthracyclines, |
| | or with mediastinal irradiation may be at higher risk. |

Plus G-CSF (see section 7.1)

#### 7.4 Transplant 1

| | Paclitaxel (Taxol) |
|---|---|
| Frequency | Toxicity |
| Common | Nausea and vomiting |
| | • Diarrhea |
| | • Mucositis |
| | • Alopecia |
| Uncommon | <ul> <li>Hypersensitivity reactions characterized by generalized skin rash, flushing, erythema, hypotension, dyspnea, and/or bronchospasm. Usually occurs within the first 2 – 10 minutes of infusion and is decreased by pre-meds</li> <li>Transient Bradycardia</li> <li>Peripheral Neuropathy - generally numbness and paresthesias</li> </ul> |
| Rare | <ul> <li>Arrythmias including Mobitz I, Mobitz II, 3<sup>rd</sup> degree heart block, and Ventricular arrhythmias</li> <li>Motor and autonomic neuropathies</li> </ul> |

| Ifosphamide (Ifex) | |
|---|---|
| Frequency | Toxicity |
| Common | <ul> <li>Nausea and vomiting with associated anorexia. An aggressive anti-emetic regimen should be used including prophylactic serotonin antagonists plus dexamethasone prior to infusion.</li> <li>Alopecia usually reversible but changes in hair color or texture after regrowth may occur</li> </ul> |
| Uncommon | • Hemorrhagic cystitis may occur despite aggressive fluid replacement, frequent voiding, and Mesna |
| Rare | • Neurotoxicity including lethargy, confusion, weakness and hallucinations may occur. This is more common in patients with impaired renal function |

#### Plus G-CSF (see section 7.1)

#### 7.5 Transplant 2

| Carboplatin (Paraplatin) | |
|---|---|
| Frequency | Toxicity |
| Common | Nausea and vomiting |
| | Hypocalcemia |
| | Hypokalemia |
| | Hypomagnesemia |
| Uncommon | Peripheral neuropathy |
| | Hyponatremia |
| | Renal toxicity |
| Rare | • Allergic reaction with infusion presenting as a skin rash, |
| | urticaria (hives), and pruritis (itching) |

| Thiotepa (Thioplex) | |
|---|---|
| Frequency | Toxicity |
| Common | Nausea and vomiting |
| | Mucositis |
| | • Skin changes including rash, bronzing of the skin, |
| | erythema, flaking, and desquamation |
| Uncommon | <ul> <li>Allergic reaction including skin rash, hives, and rarely</li> </ul> |
| | bronchospasm |
| Rare | Hemorrhagic cystitis |

| Etoposide (VP-16) | |
|---|---|
| Frequency | Toxicity |
| Common | Nausea and vomiting |
| | Diarrhea |
| | Mucositis |
| Uncommon | Hypersensitivity reaction with chills and fever |
| Rare | Bronchospasm during infusion |
| | Hypotension (low blood pressure) during infusion |

#### 7.6 Myelosuppression

7.6.1 Both the chemomobilization and the pre-transplant conditioning (chemotherapy) induce significant myelosuppression requiring re-

- infusion of viable hematopoietic stem cells for prompt hematologic recovery.
- 7.6.2 During the period of pancytopenia, the patient is highly vulnerable to infection and/or bleeding. Irradiated red cell transfusions will be given to maintain adequate oxygen delivery (hemoglobin > 8.0 gm/dL) and platelet transfusions will be given in an attempt to maintain a platelet count >10 x 10<sup>9</sup>/L.
- 7.6.3 Prophylactic measures to reduce risks of infection and to vigorously treat any infections will also be required according to UMMC BMT ID guidelines.

#### 7.7 Second malignancy

The potential carcinogenic effects of the pre-transplant chemotherapy and may compound the inherent risks of second malignancy already induced by treatment the patient may have already received. Both late second epithelial malignancies and early treatment-associated neoplasms (particularly myelodysplastic syndrome and/or leukemia) may develop after transplantation.

#### **8 Adverse Event Reporting**

Toxicity and adverse events will be classified according to NCI's Common Terminology Criteria for Adverse Events V 4.0 (CTCAE). A copy of the CTCAE can be downloaded from the CTEP home page (<a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>).

#### 8.1 Reporting Requirements

For the purposes of this study, all subjects will be monitored at least monthly continuously for all serious unexpected and selected serious adverse events (SAE) during the first 100 days after cell infusion. SAEs include: graft failure (severe pancytopenia with a marrow cellularity <5% at day +28 post transplant), relapse, and death.

Toxicities, complications of therapy and other adverse events, which are considered expected as part of therapy in general, are listed in section 7 of the protocol.

In the event of an adverse event, the first concern will be for the safety of the subject. Investigators are required to contact the PI (Dr. Claudio Brunstein,) to discuss the event and subject care.

| ADVERSE EVENT REPORTING REQUIREMENTS | | | |
|---|---|---|---|
| Unexpec | ted Event* | Expected Event* | |
| During first 100 | After first 100 | During first 100 | After first 100 days |
| days; grades 3 - 5 | days; only death or | days; selected | |
| | selected SAE** | SAE** | |
| Report using | Report using | Report using | Knowledge of Death |
| UMCC SAE form | UMCC SAE form | UMCC SAE form | and relapse reported |
| | | | annually as part of |
| | | | study continuing |
| | | | review |

<sup>\*</sup> Unexpected Events are any toxicities, complications of therapy, and adverse events NOT appearing in the Transplant Related Toxicities and Complications Section 7 of protocol.

Events that meet the reporting requirements should be simultaneously reported to the IRB and the Clinical Trials Office (CTO) within 10 working days.

The University of Minnesota Serious Adverse Event Report form may be downloaded from http://www.cancer.umn.edu/page/docs/sae.pdf

#### 9 Data and Safety Monitoring

This study will be in compliance with the University of Minnesota Cancer Center's Data & Safety Monitoring Plan, which can be accessed at http://www.cancer.umn.edu/page/resource/dataplan.html

Regular meetings of the study's principal investigator and staff will be held to discuss matters related to the safety of protocol participants, validity and integrity of the data, enrollment rate, retention of participants, adherence to protocol, and data completeness.

The Principal Investigator will provide at least monthly monitoring of patient safety with attention to the stopping rules (section 10.5) with quarterly reporting to the Clinical Trials Office (CTO) for distribution to the Data and Safety Monitoring Council (DSMC).

At the time of the IRB continuing review, the Principal Investigator will submit to the CPRC a copy of all documentation submitted to the IRB for continuing review.

<sup>\*\*</sup> Serious adverse events include: graft failure (severe pancytopenia with a marrow cellularity <5% at day +28 post transplant), relapse, and death.

#### 10 Experimental Design and Statistical Considerations

# 10.1 Primary Clinical Endpoint: Probability of one year survival for tandem AuSCT

#### 10.2 Secondary Endpoints and Comparisons

- 10.2.1 Probability of one year disease-free survival for tandem AuSCT
- 10.2.2 Toxicity rate of tandem AuSCT
- 10.2.3 Probability of engraftment of neutrophils and platelets
- 10.2.4 Determine numbers of patients unable to adequately mobilize sufficient peripheral blood stem cells (PBSC) for tandem transplant
- 10.2.5 Identify prognostic factors of those patients unlikely to mobilize sufficient PBSC for tandem transplant
- 10.2.6 Compare outcomes of overall and disease free survival for patients undergoing single versus tandem transplant due to biologic randomization

#### 10.3 Statistical Analysis

Survival and disease-free survival will be estimated by the Kaplan-Meier method. Engraftment will be estimated by cumulative incidence using competing risk methods. 95% confidence intervals will be used to make inferences. Comparison of survival and disease free survival between patients receiving single versus tandem transplant will be completed by the log-rank test or left descriptive depending on patient numbers. The toxicity rate and analysis of prognostic factors will be descriptive using proportions.

#### **10.4** Sample Size Considerations

We only expect to enroll 2 to 4 patients per year over a five year period based on a SEER incidence rate of testicular cancer in 2003 of 5.3/100,000 with a higher incidence in Caucasians, our predominant population. Since AuSCT is considered a standard salvage therapy for relapsed GCT, these patients will be seen in our clinic and most will be anticipated eligible for this study. 50-60% of patients are expected to receive a tandem AuSCT. Assuming that we enroll the maximum number of 25, we will then have 15 patients among the tandem patients to get an estimate of the survival. Assuming a survival estimate of 0.5, the 95% confidence bandwidth will have a width of 0.5.

#### 10.5 Stopping Rules

Monitoring guidelines for non-relapse mortality were developed using the sequential probability ratio test with the level of significance and power preset at 5% and 80% respectively. Monitoring guidelines will only be used for the tandem

AuSCT as single transplants have been shown to be safe in terms of non-relapse mortality.

#### Day 100 non-relapse mortality

Given a hypothesized non-relapse mortality rate of less than 5% and a maximum tolerated level of 15% among the tandem AuSCT, the trial will be halted and reviewed if 3 deaths occur in the 1<sup>st</sup> 3 evaluable patients, 5 deaths occur in the 1<sup>st</sup> 8 evaluable patients or 6 occur in the 1<sup>st</sup> 15 evaluable patients.

#### 11 Retention of Records

The investigator will retain study records, including source data, copies of case report form, study drug receipt and dispensation, and all study correspondence indefinitely in a secured facility. In addition, the Clinical Trials Office (CTO) will keep a master log of all patients participating in the study, with sufficient information to allow retrieval of the medical records for that patient.

Research data is collected in the BMT database indefinitely.

#### 12 References

- 1. Loehrer PJ, TE Ahlering, A Pollack. Testicular Cancer. In: Pazdur R, LR Coia, WJ Hoskins, LD Wagman, ed. Cancer Management: A Multidisciplinary Approach (ed 9th Edition). New York: The Oncology Group; 2005:407 -428.
- 2. International Germ Cell Consensus Classification: a prognostic factor-based staging system for metastatic germ cell cancers. International Germ Cell Cancer Collaborative Group. J Clin Oncol. 1997;15:594-603.
- 3. Bhatia S, Abonour R, Porcu P, et al. High-dose chemotherapy as initial salvage chemotherapy in patients with relapsed testicular cancer. J Clin Oncol. 2000;18:3346-3351.
- 4. Lotz JP, Bui B, Gomez F, et al. Sequential high-dose chemotherapy protocol for relapsed poor prognosis germ cell tumors combining two mobilization and cytoreductive treatments followed by three high-dose chemotherapy regimens supported by autologous stem cell transplantation. Results of the phase II multicentric TAXIF trial. Ann Oncol. 2005;16:411-418.
- 5. Mandanas RA, Saez RA, Epstein RB, Confer DL, Selby GB. Long-term results of autologous marrow transplantation for relapsed or refractory male or female germ cell tumors. Bone Marrow Transplant. 1998;21:569-576.
- 6. Nichols CR, Andersen J, Lazarus HM, et al. High-dose carboplatin and etoposide with autologous bone marrow transplantation in refractory germ cell cancer: an Eastern Cooperative Oncology Group protocol. J Clin Oncol. 1992;10:558-563.

- 7. Beyer J, Kramar A, Mandanas R, et al. High-dose chemotherapy as salvage treatment in germ cell tumors: a multivariate analysis of prognostic variables. J Clin Oncol. 1996;14:2638-2645.
- 8. Attal M, Harousseau JL, Facon T, et al. Single versus double autologous stem-cell transplantation for multiple myeloma. N Engl J Med. 2003;349:2495-2502.
- 9. Margolin BK, Doroshow JH, Ahn C, et al. Treatment of germ cell cancer with two cycles of high-dose ifosfamide, carboplatin, and etoposide with autologous stem-cell support. J Clin Oncol. 1996;14:2631-2637.
- 10. Motzer RJ, Mazumdar M, Sheinfeld J, et al. Sequential dose-intensive paclitaxel, ifosfamide, carboplatin, and etoposide salvage therapy for germ cell tumor patients. J Clin Oncol. 2000;18:1173-1180.
- 11. Margolin KA, Doroshow JH, Frankel P, et al. Paclitaxel-based high-dose chemotherapy with autologous stem cell rescue for relapsed germ cell cancer. Biol Blood Marrow Transplant. 2005;11:903-911.
- 12. Chou TC, Motzer RJ, Tong Y, Bosl GJ. Computerized quantitation of synergism and antagonism of taxol, topotecan, and cisplatin against human teratocarcinoma cell growth: a rational approach to clinical protocol design. J Natl Cancer Inst. 1994;86:1517-1524.
- 13. Kollmannsberger C, Nichols C, Bokemeyer C. Recent advances in management of patients with platinum-refractory testicular germ cell tumors. Cancer. 2006;106:1217-1226.
- 14. Motzer RJ, Bajorin DF, Schwartz LH, et al. Phase II trial of paclitaxel shows antitumor activity in patients with previously treated germ cell tumors. J Clin Oncol. 1994;12:2277-2283.
- 15. Vaena DA, Abonour R, Einhorn LH. Long-term survival after high-dose salvage chemotherapy for germ cell malignancies with adverse prognostic variables. J Clin Oncol. 2003;21:4100-4104.
- 16. Rick O, Bokemeyer C, Beyer J, et al. Salvage treatment with paclitaxel, ifosfamide, and cisplatin plus high-dose carboplatin, etoposide, and thiotepa followed by autologous stem-cell rescue in patients with relapsed or refractory germ cell cancer. J Clin Oncol. 2001;19:81-88.
- 17. Motzer RJ, Mazumdar M, Bosl GJ, Bajorin DF, Amsterdam A, Vlamis V. High-dose carboplatin, etoposide, and cyclophosphamide for patients with refractory germ cell tumors: treatment results and prognostic factors for survival and toxicity. J Clin Oncol. 1996;14:1098-1105.
- 18. Rosti G, De Giorgi U, Salvioni R, et al. Salvage high-dose chemotherapy in patients with germ cell tumors: an Italian experience with 84 patients. Cancer. 2002;95:309-315.

# **Appendix I: International Germ Cell Cancer Consensus Classification**

| Non-Seminomas | SEMINOMAS |
|---|---|
| Good Pro | gnosis |
| Testicular or retroperitoneal primary <u>AND</u> | Any primary site <u>AND</u> |
| <ul> <li>No non-pulmonary visceral metastases <u>AND</u></li> </ul> | No non-pulmonary visceral metastases |
| <ul> <li>Good Markers defined as (requires all)</li> </ul> | AND |
| AFP < 1000 ng/mL | Markers |
| hCG < 5000 IU/L | AFP: normal |
| LDH < 1.5 x Upper limit of normal | hCG and LDH: normal or elevated |
| <b>Intermediate</b> | Prognosis |
| Testicular or retroperitoneal primary <u>AND</u> | Any primary site <u>AND</u> |
| <ul> <li>No non-pulmonary visceral metastases <u>AND</u></li> </ul> | <ul> <li>Non-pulmonary visceral metastases <u>AND</u></li> </ul> |
| <ul> <li>Intermediate Markers defined as any of</li> </ul> | Markers |
| AFP 1000 – 10,000 ng/mL | AFP: normal |
| hCG 5000 – 50,000 IU/L | hCG and LDH: normal or elevated |
| LDH 1.5 – 10 x Upper limit of normal | |
| Poor Prog | gnosis |
| <ul> <li>Mediastinal primary <u>OR</u></li> </ul> | No patients with pure seminomas are |
| <ul> <li>Non-pulmonary visceral metastases <u>OR</u></li> </ul> | classified as poor prognosis |
| <ul> <li>Poor Markers defined as any of</li> </ul> | |
| AFP > 10,000 ng/mL | |
| hCG > 50,000 IU/L | |
| LDH > 10 x Upper limit of normal | |

# **Appendix II – Lansky and Karnofsky Performance Status**

| LANSKY (persons < 16 years old) | | KARNOFSKY (persons ≥ 16 years old) |
|---|---|---|
| Fully active, normal | 100 | Normal no complaints; no evidence of disease. |
| Minor restrictions in physically strenuous activity | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| Active, but tires more quickly | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Both greater restriction of and less time spent in play activity | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| Up and around, but minimal active play; keeps busy with quieter activities | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| Gets dressed but lies around much of the day, no active play but able to participate in all quiet play and activities | 50 | Requires considerable assistance and frequent medical care. |
| Mostly in bed; participates in quiet activities | 40 | Disabled; requires special care and assistance. |
| In bed; needs assistance even for quiet play | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| Often sleeping; play entirely limited to very passive activities | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| No play; does not get out of bed | 10 | Moribund; fatal processes progressing rapidly. |
| Unresponsive | 0 | Dead |

Appendix IIIA: Required Observations <u>Transplant 1</u>

| | within 30<br>days of<br>enrollment | Prior to<br>Admit for<br>transplant | day<br>+14 | day<br>+28 | day +42 | day +60 | day +74 | day +88 | **<br>day<br>+100 | day<br>+180 | 9 mo | 1 yr | 18 mo | 2yr |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Medical History | X | х | | | | | | | | | | | | |
| Physicial Exam | X | Х | | X | | Х | | | X | Х | | х | X | Х |
| Weight/Height | X | X | | | | | | | | | | | | |
| Performance status | X | X | | X | | X | | | X | Х | | X | X | X |
| Adverse Event/toxicity notation | X | X | | X | | х | | | X | X | | X | X | X |
| Comprehensive chemistry panel | X | X | | X | | х | | | X | X | | X | X | Х |
| Hepatic Panel | X | X | | X | | х | | | X | X | | X | X | Х |
| CBC with diff | X | X | | X | | X | | | X | Х | | X | X | X |
| AFP | X | X | X | X | X | X | X | Х | X | Х | X | X | X | X |
| LDH | X | X | X | X | X | х | х | Х | X | X | X | X | X | Х |
| β-hCG | X | X | X | X | X | X | X | Х | X | Х | X | X | X | X |
| Viral Hepatitis serologies | X | | | | | | | | | | | X | | |
| Quantitative Immunoglobulin | X | | | | | | | | X | X | | X | | |
| pb CD4 <sup>+</sup> | X | | | | | | | | X | X | | X | | |
| pb CD8 <sup>+</sup> | X | | | | | | | | X | X | | X | | |
| CT scan – chest, abdomen, pelvis, and head. PET/CT will be done at all timepoints except d+28. | x | | | X | | | | | X | X | | x | X | X |
| Bone Scan | X | | | | | | | | | X | | х | X | X |
| MRI brain (if prior CNS lesions) | X | | | X | | | | | X | | | х | | |
| Bilateral bm biopsy unilateral aspirate | X | | | | | | | | | | | х | | X |
| BM Cytogenetics | X | | | | | | | | | | | X | | X |

An attempt should be made to obtain the scheduled activity as close as possible to the scheduled date. However, scheduling difficulties (for procedures and around weekends) may make this difficult. Therefore, the scheduled activity will be obtained within 14 days of that schedule (30 days for dates after day +100).

\*\*For patients NOT having a second transplant, all follow-up procedures will continue out to 2 years based on the Required Observations table for <u>Transplant 1</u>. For patients having a second transplant, required observations will be per the Required Observations table for Transplant 2 and no further Transplant 1 observations will be collected.

7/12/2019 

Appendix IIIB: Required Observations <u>Transplant 2</u> (This will start between day +30 and day +90 from transplant 1)

| | Within 2 wks<br>of planned<br>admission | day<br>+14 | day<br>+28 | day +42 | day +60 | day +74 | day +88 | day<br>+100 | day<br>+180 | 9 mo | 1 yr | 18 mo | 2yr |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Medical History | х | | | | | | | | | | | | |
| Physicial Exam | X | | X | | X | | | X | X | | x | X | X |
| Weight/Height | X | | | | | | | | | | | | |
| Performance status | X | | X | | X | | | X | X | | х | X | X |
| Adverse Event/toxicity notation | X | | X | | X | | | X | X | | X | X | X |
| Comprehensive chemistry panel | X | | X | | X | | | X | X | | x | X | X |
| Hepatic Panel | X | | X | | X | | | X | X | | x | X | X |
| CBC with diff | X | | X | | X | | | X | X | | x | X | X |
| AFP | X | X | X | х | X | Х | X | X | X | X | x | X | X |
| LDH | X | X | X | х | X | Х | X | X | X | X | x | X | X |
| β-hСG | X | X | X | х | X | Х | X | X | X | X | x | X | X |
| Viral Hepatitis serologies | X | | | | | | | | | | х | | |
| Quantitative Immunoglobulin | X | | | | | | | X | X | | X | | |
| pb CD4 <sup>+</sup> | X | | | | | | | X | X | | X | | |
| pb CD8 <sup>+</sup> | X | | | | | | | X | X | | x | | |
| CT scan – chest, abdomen, pelvis, and head. PET/CT will be done at all timepoints except d+28. | x | | X | | | | | х | X | | X | X | х |
| Bone Scan | | | | | | | | | X | | X | X | х |
| MRI brain (if prior CNS lesions) | X | | X | | | | | X | | | X | | |
| Bilateral bm biopsy unilateral aspirate | | | | | | | | | | | X | | X |
| BM Cytogenetics | | | | | | | | | | | х | | X |

An attempt should be made to obtain the scheduled activity as close as possible to the scheduled date. However, scheduling difficulties (for procedures and around weekends) may make this difficult. Therefore, the scheduled activity will be obtained within 14 days of that schedule (30 days for dates after day +100).

7/12/2019 

APPENDIX IV: RECIST Criteria

#### Response Criteria

#### **Evaluation of target lesions \***

Complete Response (CR): Disappearance of all target lesions

Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking

as reference the baseline sum LD

Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the

smallest sum LD recorded since the treatment started or the appearance of one or

more new lesions

Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD,

taking as reference the smallest sum LD since the treatment started

**Evaluation of non-target lesions** 

Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor marker level

Incomplete Response/
Persistence of one or more non-target lesion(s) or/and maintenance of tumor marker

Stable Disease (SD): level above the normal limits

Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing

non-target lesions \*\*

<sup>\*</sup> Target lesions: any lesion measurable prior to therapy. Lesions must be  $\geq 1$  cm in longest diameter at time of disease evaluation prior to autologous transplant.

<sup>\*\*</sup>Although a clear progression of "non target" lesions only is exceptional, in such circumstances, the opinion of the treating physician should prevail and the progression status should be confirmed later on by the review panel (or study chair).